CLINICAL TRIAL: NCT03054051
Title: A Mobile Phone Game to Prevent HIV Among Young Africans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Kate Winskell, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00081150; 5R34MH106368 (NIH)
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Results first posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-09

CONDITIONS: HIV/AIDS
Keywords: HIV prevention; Preadolescence; Mobile phone game; Feasibility
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumaini Mobile Phone Game (Experimental): Participants randomized to this arm will be invited to play the Tumaini game.
  Interventions: Behavioral: Tumaini Mobile Phone Game
- Standard of Care (No Intervention): Participants randomized to this arm will receive no intervention beyond the current standard of care for sexual education.

INTERVENTIONS:
Behavioral: Tumaini Mobile Phone Game — Tumaini is a scenario-based role-playing game application, optimized for use on low-cost Android smartphones. Participants will be invited to play the game for at least ten hours over a period of three weeks. The game is designed to: educate players about sexual health and HIV/AIDS; build risk-reduction skills and related self-efficacy for prevention of HIV/STIs and unintended pregnancy; challenge HIV stigma and harmful gender norms; and promote parent-child dialogue.
  Arms: Tumaini Mobile Phone Game

SUMMARY:
This project will test the feasibility of an electronic game to prevent HIV among African preadolescents, delivered via inexpensive Android smart phones. In order to collect feasibility data for a future randomized controlled trial, this study involves the pilot-testing of the intervention with a sample of young people in Nyanza region, Kenya, where 11.4% of young women ages 15-24 are HIV-infected. This feasibility study will be carried out with the Kenya Medical Research Institute (KEMRI).

DETAILED DESCRIPTION:
This project will test the feasibility of an electronic game for preadolescents, delivered via inexpensive Android smart phones. The game is informed by socio-behavioral and pedagogical theories, evidence-based practice, and formative research on youth sexual culture in sub-Saharan Africa. It is designed to: educate young players, ages 11-14, about sexual health and HIV/AIDS; build risk-reduction skills and related self-efficacy for prevention of HIV, sexually transmitted infections (STIs), and unintended pregnancy; challenge harmful gender norms and HIV stigma; and foster dialogue with parents and caregivers.

The proposed feasibility test will be conducted in Western Kenya. Sixty preadolescents will be enrolled in the trial, 30 in the study arm and 30 in the control arm. The Kenya Medical Research Institute (KEMRI) has established community advisory boards (CABs) in Kisumu, which will be available to the proposed study.

Data collection will take place at KEMRI offices, health clinics, or in the meeting room of a local community-based organization (CBO). In addition, data on game-play will be automatically collected on mobile phones given to preadolescent study participants.

ELIGIBILITY:
Inclusion criteria:

* Aged 11-14 at time of recruitment
* Resident in Nyanza region, Kenya
* Having basic literacy in English
* Only one child enrolled per family

Exclusion criteria:

* Aged <11 or >14 at time of recruitment
* Not resident in Nyanza region, Kenya
* Without basic literacy in English
* Sibling to a child already enrolled in the study
* Participant in formative research to inform the study

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Winskell, PhD, Principal Investigator — Emory University
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Winskell K, Sabben G, Akelo V, Ondeng'e K, Obong'o C, Stephenson R, Warhol D, Mudhune V. A Smartphone Game-Based Intervention (Tumaini) to Prevent HIV Among Young Africans: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Aug 1;6(8):e10482. doi: 10.2196/10482. PMID 30068501
- [Result] Sabben G, Akelo V, Mudhune V, Ondeng'e K, Ndivo R, Stephenson R, Winskell K. A Smartphone Game to Prevent HIV Among Young Africans: Protocol for a Randomized Pilot Study of a Mobile Intervention. JMIR Res Protoc. 2019 Mar 27;8(3):e11209. doi: 10.2196/11209. PMID 30916661
- [Result] Sabben G, Mudhune V, Ondeng'e K, Odero I, Ndivo R, Akelo V, Winskell K. A Smartphone Game to Prevent HIV Among Young Africans (Tumaini): Assessing Intervention and Study Acceptability Among Adolescents and Their Parents in a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 May 21;7(5):e13049. doi: 10.2196/13049. PMID 31115348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from schools in Kisumu Town, western Kenya, Africa. Enrollment of participants occurred between March 20, 2017 and April 7, 2017. All study activities were completed by June 19, 2017.
Pre-assignment Details: Letters were sent to 150 parent of age-eligible children inviting them to attend informational meetings. Of the 126 who attended a meeting, 90 were interested and eligible to participate and 60 of these were randomly selected to enroll in the study.
Groups:
- Tumaini Mobile Phone Game: Participants randomized to this arm were invited to play the Tumaini game. Participants were asked to play the game for at least one hour per day for 16 days.
- Standard of Care: Participants randomized to this arm received no intervention beyond the current standard of care for sexual education.
Period: Overall Study
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tumaini Mobile Phone Game | Standard of Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (1) | 12.6 (1) | 12.7 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 16 | 14 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number Interested in Participating
Description: To evaluate the feasibility of conducting a technology based intervention in a low resource area, the number of eligible individuals who were interested in participating after hearing about the study was examined. Letters were sent to 150 families inviting them to attend an informational meeting and 126 attended a meeting and were assess for eligibility.
Time Frame: Month 1
Population: This analysis includes all of the individuals who expressed interest in the study by attending an informational meeting.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Study participants who were randomized to either the intervention or control arm.
Arm/Group | All Study Participants
Number analyzed (Participants) | 126
Participants
  Uninterested | 2
  Did not meet inclusion criteria | 34
  Eligible and interested | 90

2. Primary Outcome: Time to Recruitment of 60 Participants
Description: The number of days needed to recruit 60 participants.
Time Frame: Month 1
Measure: Number; unit: days
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
days | 18

3. Primary Outcome: Number of Participants Lost to Follow Up
Description: The number of participants who consented to participate but then later could not be reached prior to completing all study visits.
Time Frame: Duration of Study (Up to 4 Months)
Measure: Count of Participants; unit: Participants
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

4. Primary Outcome: Number of Participants Completing the Study
Description: The number of participants who completed all study visits after providing consent are presented here.
Time Frame: Duration of Study (Up to 4 Months)
Measure: Count of Participants; unit: Participants
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Number analyzed (Participants) | 30 | 30
Participants | 30 | 30

5. Primary Outcome: Number of Phones Returned
Description: The phone retention rate (phones not lost during the intervention) was assessed by the number of phones returned at the end of the intervention.
Time Frame: Month 2
Measure: Number; unit: phones
Groups:
- Tumaini Mobile Phone Game: Participants randomized to this arm were invited to play the Tumaini game.
Arm/Group | Tumaini Mobile Phone Game
Number analyzed (Participants) | 30
phones | 30

6. Primary Outcome: Number Reporting Game Was Very Fun
Description: Game acceptability was assessed by asking participants how fun playing the game was. The number of participants reporting that the game was "very fun" are presented here.
Time Frame: Day 17 (post-intervention)
Population: This analysis includes participants in the intervention arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tumaini Mobile Phone Game
Number analyzed (Participants) | 30
Participants | 27

7. Primary Outcome: Number Reporting the Game is Valuable
Description: The value of the game was assessed with several questions regarding how much the participants learned and how useful the information is. The number of participants reporting that they learned a lot, found the information very useful now, and found the information very useful for the future, are presented below.
Time Frame: Day 17 (post-intervention)
Population: This analysis includes participants randomized to the intervention arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tumaini Mobile Phone Game
Number analyzed (Participants) | 30
Participants
  Learned A Lot | 30
  Information Very Useful Now | 29
  Information Very Useful for Future | 30

8. Primary Outcome: Number of Participants Feeling Very Safe
Description: Personal safety associated with being in possession of the phone was assessed by the post-intervention survey. Phones provided for the intervention were set up so that all other features were blocked and only function the phone could perform was playing the game.
Time Frame: Day 17 (post-intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Tumaini Mobile Phone Game
Number analyzed (Participants) | 30
Participants | 29

9. Primary Outcome: Number of Participants Playing the Game
Description: Participants were asked to play the game for at least one hour per day for 16 days. The number of participants who reported playing the game everyday and the number of participants who reported playing the game for an hour or more each time are presented here.
Time Frame: Day 17 (post-intervention)
Population: Only participants randomized to the intervention arm are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tumaini Mobile Phone Game
Number analyzed (Participants) | 30
Participants
  Reported played every day | 26
  Reported played 1 hour or more every time | 23

10. Secondary Outcome: Change in Knowledge
Description: Knowledge measures will be assessed via Yes/No survey questions and will address puberty, HIV, sexually transmitted infections (STIs), pregnancy, condoms, and alcohol and drugs. Knowledge was assessed with 15 items and responses are coded as 0 or 1. Total scores range from 0 to 15, with higher scores indicating increased knowledge. A positive value for the change from baseline score indicates an increase in knowledge from the baseline assessment.
Time Frame: Baseline, Day 17 (post-intervention), 6 Weeks Post-intervention
Population: One participant from the intervention arm was removed from this analysis at the immediate post-intervention time point due to delayed completion of the post-intervention survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline score | 7.33 (2.12) | 7.93 (1.74)
  Change from baseline immediately post-intervention: number analyzed (Participants) | 29 | 30
  Change from baseline immediately post-intervention | 4.76 (2.96) | 0.27 (2.07)
  Change from baseline at 6 weeks post-intervention | 3.80 (2.37) | 0.80 (2.14)

11. Secondary Outcome: Change in Self-Efficacy
Description: Self-efficacy was assessed via a 3-point Likert scale, and addressed self-efficacy to seek advice about puberty, sex, relationships; to communicate about protected sex; to reject peer, partner and adult pressure to engage in risk behaviors. Self-efficacy was assessed with 9 items which were scored as 0, 0.5 or 1. Total scores ranged from 0 to 9, with higher scores indicating increased self-efficacy. A positive value for the change from baseline score indicates an increase in self-efficacy since the baseline assessment.
Time Frame: Baseline, Day 17 (post-intervention), 6 Weeks Post-intervention
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline score | 5.87 (2.03) | 6.22 (2.41)
  Change from baseline immediately post-intervention: number analyzed (Participants) | 29 | 30
  Change from baseline immediately post-intervention | 1.95 (1.57) | 0.47 (1.07)
  Change from baseline at 6 weeks post-intervention | 2.03 (1.83) | 0.63 (1.20)

12. Secondary Outcome: Change in Risk Assessment
Description: Risk assessment was assessed via a 3-point Likert scale, and addressed perceived risk of certain risk situations/behaviors and of contracting HIV. Risk is assessed with 4 items and responses are coded as 0, 0.5 or 1. Total scores range from 0 to 4, with higher scores indicating increased risk assessment. A positive value for the change from baseline score indicates an increase in assessing risky situations as risky.
Time Frame: Baseline, Day 17 (post-intervention), 6 Weeks Post-intervention
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline score | 2.67 (1.25) | 2.45 (1.50)
  Change from baseline immediately post-intervention: number analyzed (Participants) | 29 | 30
  Change from baseline immediately post-intervention | 0.41 (1.17) | 0.00 (1.23)
  Change from baseline at 6 weeks post-intervention | 0.52 (0.99) | 0.07 (1.03)

13. Secondary Outcome: Change in Behavioral Intention
Description: Behavioral intention was assessed via Yes/No questions. The measure addressed intention to seek advice, to avoid risk situations, and to engage in health protective behaviors. Behavioral intention is assessed with 6 items that are scored as 0 or 1 and total scores range from 0 to 6. Higher scores in indicate more intention to partake in health protective behaviors and a positive value for the change from baseline score indicates a desirable change in intention.
Time Frame: Baseline, Day 17 (post-intervention), 6 Weeks Post-intervention
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline score | 4.43 (0.77) | 4.83 (0.70)
  Change from baseline immediately post-intervention: number analyzed (Participants) | 29 | 30
  Change from baseline immediately post-intervention | 0.28 (0.86) | -0.12 (0.76)
  Change from baseline at 6 weeks post-intervention | 0.43 (0.75) | -0.15 (0.82)

14. Secondary Outcome: Change in Future Orientation
Description: Future orientation was assessed via a single multiple-choice question (Yes/No/Maybe) and addressed perceived locus of control. Response is coded as 0, 0.5, or 1 and higher scores indicate greater understanding of future locus of control. A positive value for the change from baseline score indicates a desirable change in scores.
Time Frame: Baseline, Day 17 (post-intervention), 6 Weeks Post-intervention
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline score | 0.86 (0.30) | 0.90 (0.24)
  Change from baseline immediately post-intervention: number analyzed (Participants) | 29 | 30
  Change from baseline immediately post-intervention | 0.05 (0.34) | 0.10 (0.34)
  Change from baseline at 6 weeks post-intervention | 0.04 (0.31) | 0.08 (0.27)

15. Secondary Outcome: Change in Perceived Social Norms
Description: Perceived social norms were assessed via a 3-point Likert and addressed sex, gender, condoms, and HIV stigma. Social norms were assessed with 6 items that are scored as 0, 0.5, or 1. Total scores range from 0 to 6 with higher scores indicating perception of more desirable social norms. A positive value for the change from baseline scores indicates a desirable change.
Time Frame: Baseline, Day 17 (post-intervention), 6 Weeks Post-intervention
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline score | 3.72 (1.12) | 3.67 (1.24)
  Change from baseline immediately post-intervention: number analyzed (Participants) | 29 | 30
  Change from baseline immediately post-intervention | 0.47 (1.26) | -0.07 (1.30)
  Change from baseline at 6 weeks post-intervention | 0.37 (0.37) | -0.15 (1.35)

16. Secondary Outcome: Change in Attitudes
Description: Attitudes were assessed via 3-pt Likert survey questions relating to HIV stigma, condoms, sex, gender, and future orientation. Attitudes were assessed with 15 items and responses coded as 0, 0.5, or 1. Total scores ranged from 0 to 15, with higher scores indicating more desirable attitudes. A positive value for the change from baseline score indicates an increase in desirable attitudes.
Time Frame: Baseline, Day 17 (post-intervention), 6 Weeks Post-intervention
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline score | 9.95 (2.30) | 9.22 (2.07)
  Change from baseline immediately post-intervention: number analyzed (Participants) | 29 | 30
  Change from baseline immediately post-intervention | 0.74 (2.13) | 0.82 (1.95)
  Change from baseline at 6 weeks post-intervention | 1.18 (1.82) | 0.80 (2.25)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time participants signed the consent form through the 6 week post-intervention study visit.
Arm/Group | Tumaini Mobile Phone Game | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03054051/Prot_SAP_ICF_000.pdf